CLINICAL TRIAL: NCT06676111
Title: The Effectiveness of Probiotics in Relieving Allergic Rhinitis in Children and Their Regulatory Effect on the Gut Microbiota and Metabolic Profile
Brief Title: Effectiveness of Probiotics in Relieving Allergic Rhinitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024009
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Children With Allergic Rhinitis
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Probiotic pectin gummies(2 billion CFU)/2 pellets/day BC99; Storage: Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): No probiotic pectin gummies/2 pellets/day; Storage: Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study lasts 56 days and each patient will have 3 visits (W0, W4, W8)
  Arms: Probiotic group
Dietary Supplement: Placebo — The experimental phase of this study lasts 56 days and each patient will have 3 visits (W0, W4, W8)
  Arms: Placebo group

SUMMARY:
To evaluate the clinical efficacy of probiotic gummies in the trial of allergic rhinitis in children compared to placebo, as well as the modulating effect on gut microbiota, serum metabolic profile, and occurrence of adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary, written, and signed informed consent form, agreeing to participate in this study;
2. Capable of completing research according to the requirements of the experimental plan;
3. Age range: 4-14 years old;
4. Meets the diagnostic criteria for AR established in the "Guidelines for Diagnosis and Treatment of Allergic Rhinitis in Children (Revised 2022)";
5. Symptoms: Two or more symptoms appear: sneezing, watery nasal discharge, nasal itching, and nasal congestion. Symptoms last or accumulate for more than 1 hour per day, and may be accompanied by eye symptoms such as itching, tearing, and redness;
6. Physical signs: pale and edematous nasal mucosa, accompanied by watery discharge.

Exclusion Criteria:

1. Drugs that affect the intestinal flora (including antibacterial drugs, probiotics, intestinal mucosal protective agents, traditional Chinese patent medicines and simple preparations, etc.) are continuously used for more than one week within one month before screening;
2. Merge with tuberculosis patients;
3. Combined with allergic asthma;
4. Patients with nasal polyps or severe nasal septum deviation;
5. Patients with serious systemic diseases or malignant tumors;
6. Individuals with congenital genetic disorders or congenital immunodeficiency diseases;
7. Regular use of probiotics or prebiotics within the first 6 months of the screening period;
8. Individuals with severe gastrointestinal diseases (including severe diarrhea, inflammatory bowel disease, etc.);
9. Those with metabolic syndrome (including obesity, abnormal lipid metabolism, hypertension, diabetes, etc.);
10. Patients with combined sinusitis, otitis media, or respiratory infections;
11. Stop taking the test sample or add other drugs midway, unable to determine efficacy or incomplete data;
12. Short term use of substances with similar functions to the test subject affects the judgment of the results;
13. The subject is unable to participate in the trial due to personal reasons;
14. Participants deemed unsuitable by other researchers to participate. Those who meet any of the above conditions shall not be selected.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score (TNSS) | 56 days
  Score 0 - asymptomatic; Score 1 - mild symptoms, easily tolerated; Score 2 - moderate symptoms, annoying but tolerable; Score 3 - Severe symptoms, intolerable, affecting daily life and sleep. Add them together to get the total score
Visual Analogue Scale (VAS) | 56 days
  "0" means no such symptoms; "10" means that this symptom is the most severe. Add them together to get the total score
Rhinoconjunctivitis-related quality of life questionnaire (RQLQ) | 56 days
  0 points: no trouble; 1 point: little to no distress; 2 points: occasional distress; Score 3: Moderate degree of distress; 4: Somewhat bothered, 5: Very bothered; Score 6: Extremely distressed
Medication scores | 56 days
  Scoring drugs include oral antihistamines (3 points/tablet, maximum 6 points), oral leukotriene receptor antagonists (2 points/dose), nasal glucocorticoids (1 point/spray, maximum 8 points), nasal spray or eye drops antihistamines (0.5 points/spray or drop, maximum 4 points), and the daily average score for the past 1 week was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Science and Technology, Luoyang, Henan, China

REFERENCES:
- [Derived] Han Z, Zhu H, Yang Y, Wang Y, Li X, Zhu J, Wu Y, Fang S, Gu S. Weizmannia coagulans BC99 alleviates pediatric allergic rhinitis via the gut microbiota-SCFAs- immunomodulatory axis: A randomized, double-blind, placebo-controlled trial. Int Immunopharmacol. 2026 Jan 1;168(Pt 1):115787. doi: 10.1016/j.intimp.2025.115787. Epub 2025 Nov 5. PMID 41197269